CLINICAL TRIAL: NCT04415476
Title: A Randomized, Open-label,Controlled Phase II b Study to Demonstrate Efficacy and Safety of Sirolimus Chronic Rejection After Lung Transplant
Brief Title: Standard Therapy Using Tacrolimus, Mycophenolate Mofetil and Prednisone For Chronic Lung Transplant Rejection (BOS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not proceed to IRB approval.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00091412
Record Dates: First submitted 2020-05-13; First posted 2020-06-04 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2020-06

CONDITIONS: Disorder Related to Lung Transplantation; Chronic Rejection of Lung Transplant; Decreased Immunologic Activity
Keywords: lung function; Lung Transplantation; case-control study; bronchiolitis obliterans syndrome (BOS)
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Tacrolimus; Mycophenolic Acid; Prednisone; Sirolimus

STUDY DESIGN:
Intervention Model Description: Paralled Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirolimus and Tacrolimus and prednisone (Other): Assigned Interventions Sirolimus (Rapamune) Tacrolimus (Prograft) Prednisone (Deltasone, Prednicot, Rayos, Sterapred)
  Interventions: Drug: Assigned Interventions
- Standard of Care (Experimental): Arm1:) sirolimus and tacrolimus and prednisone group:
  Tacrolimus, The patient will receive 0.1-0.15 mg/kg/day PO in 2 divided doses Adjust trough blood 5-12 ng/ml.
  Mycophenolate mofetil (NA )Stopped upon sirolimus initiation Sirolimus:1-5 mg/day PO if >40 kg / 1 mg/m²/day if <40 kg trough blood levels 5-12 ng/ml Prednisone:20 mg/day PO if >40 kg and 10 mg/day if <40 kg, adjust based on adverse effects.
  Arm 2) Standard Therapy Tacrolimus:0.1 to 0.15 mg/kg/day PO in 2 divided doses Adjust trough blood 8-12 ng/ml Mycophenolate mofetil:750-1250 mg bid PO and adjust to tolerance (WBCs and GI side effects Sirolimus: NA Prednisone: Prednisone dose 20 mg/day PO if >40 kg and 10 mg/day if <40 kg, adjust based on adverse effect
  Interventions: Drug: Assigned Interventions

INTERVENTIONS:
Drug: Assigned Interventions — This is a prospective single-center, open-label, randomized, controlled pilot study in the treatment of chronic rejection (CR), defined as grade 1 and 2 BOS, in adult recipients of a pulmonary allograft (single or double lungs). Patients meeting entry criteria shall demonstrate a sustained decline in FEV1 having met stage 1 or 2 BOS. Patients randomized to the study arm, will be treated with Sirolimus (S) orally in place of MMF in addition to tacrolimus and prednisone compared to those patients randomized to defined ST alone (tacrolimus, MMF and prednisone). The trial duration will be approximately 2 years for each subject randomized. Treatment compliance and safety will be monitored by clinic visits at 4-6 week intervals for the 2 year subject duration and will include standard physical examinations and monitoring of routine clinical and laboratory parameters including cause of hospitalizations and rate of adverse events including death in each group. T
  Other Names: Tacrolimus; Mycophenolate mofetil; Prednisone; Sirolimus; Prograft; Cellcept; Deltasone; Prednicot; Rayos; Sterapred; Rapamune

SUMMARY:
This is a prospective single-center, open-label, randomized, controlled pilot

study in the treatment of chronic rejection (CR), defined as grade 1 and 2

BOS, in adult recipients of a pulmonary allograft (single or double lungs).To assess the efficacy and safety of sirolimus plus tacrolimus and prednisone

(S) compared to standard therapy (tacrolimus, mycophenolate mofetil

(MMF) and prednisone) (ST) for chronic rejection, defined as grades 1 and 2

bronchiolitis obliterans syndrome (BOS); BOS defined as ≥ 20% decline

from maximal post-transplant FEV1.

DETAILED DESCRIPTION:
This is a prospective single-center, open-label, randomized, controlled pilot

study in the treatment of chronic rejection (CR), defined as grade 1 and 2

BOS, in adult recipients of a pulmonary allograft (single or double lungs).

Patients meeting entry criteria shall demonstrate a sustained decline in FEV1

having met stage 1 or 2 BOS. Patients randomized to the study arm, will be

treated with Sirolimus (S) orally in place of MMF in addition to tacrolimus

and prednisone compared to those patients randomized to defined ST alone

(tacrolimus, MMF and prednisone). The trial duration will be approximately

Primary endpoints will include:

Efficacy failure between ST and S randomized group investigational treatment regimens will be determined at 96 weeks after the last patient is randomization and enrolled at approximately study year 2. The control arm will receive standard of care treatment (ST) and immunosuppression according to the University of Maryland lung transplant protocol. Efficacy failure will be defined as the combined end point of progression of BOS (defined as at least a 20 % decline from the initial randomization FEV1 value confirmed by two separate measurements three weeks apart or more) or re-transplantation or death. The co-primary end point of FEV1 and FVC changes to define functional stabilization in the S arm compared to ST is to be completed when the last patient randomized (patient #30) has been enrolled for 2 years as well.

Efficacy of S is to be assessed using following parameters to determine its effect on lung function:

1. Forced expiratory volume in one second (FEV1)
2. Forced vital capacity (FVC)
3. FEF 25-75

Secondary endpoints will include:

* General S tolerability
* Incidence and severity of adverse events (AE)
* Changes in clinical laboratory parameters from baseline after randomization
* Changes in vital signs
* Changes in physical examinations
* Incidence of infections
* Average maintenance doses of calcineurin inhibitors, antimetabolite agents, and corticosteroids
* Number of courses of augmented immunosuppressants
* Number and days of hospitalization
* Incidence of malignancies
* Overall mortality (including transplant-related mortality)
* Retransplantation

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 or older.
2. Recipient of a single or double pulmonary allograft at least twelve months before study entry.
3. Clinically diagnosed BOS grade 1 or 2
4. Receiving oral TAC-based immunosuppression according to institutional standards.
5. Capable of understanding the purposes and risks of the study, has given written informed consent and agrees to comply with the study requirements and capable of protocol adherence.
6. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to study entry.
7. Stable to enable routine pre and post-transplant bronchoscopy with BAL and biopsy.
8. Fasting cholesterol < 250 mg/dL, fasting triglycerides < 250 mg/dL -

Exclusion Criteria:

1. Active bacterial, viral or fungal infection not successfully resolved at least 4 weeks prior to study entry.
2. Mechanical ventilation.
3. At screening FEV1 < 1 liter and/or < FEV1 of 25 % predicted.
4. Pregnant women or women who are unwilling to use appropriate birth control to avoid pregnancy.
5. Women who breastfeed.
6. Known hypersensitivity to sirolimus.
7. Serum creatinine value of > 2.5 mg/dL or chronic dialysis use or liver disease with a bilirubin > 2 mg/dL.
8. Subjects with severe underlying disease other than BOS that is thought to become fatal within four months of clinical assessment.
9. Receipt of an investigational drug as part of a clinical trial within 4 weeks prior to study entry. This is defined as any treatment that is implemented under an Investigational New Drug.
10. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary procedures.
11. Any co-existing medical condition that in the Investigator's judgment will substantially increase the risk associated with the patient's participation in the clinical trial.
12. Clinically significant bronchial strictures unresponsive to dilatation procedures.
13. Subjects with malignancy diagnosed within one year prior to screen (with the exception of skin cancers).
14. Lipid panel fasting cholesterol > 250 mg/dL, fasting triglycerides >250 mg/dL

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Death | 2 years
  Increase in motility
Re-Transplantation | 2 years
  Increase in re-transplantation from baseline
FEV1 (Forced Respiratory Volume in 1 second) | 2 years
  Greater or equal to 20% decline in FEV1 from randomization

SECONDARY OUTCOMES:
FVC (Forced Vital Capacity) | 2 years
  Caparison between the two treatment groups.
FEF (forced expiratory flow) | 2 years
  The rate of airflow recorded in measurements of forced vital capacity, usually calculated as an average flow over a given portion of the expiratory curve; the portion between 25 and 75 per cent of forced vital capacity.
  Comparison on FEF(25-75) between the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo T Iacono, MD, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iacono AT, Johnson BA, Grgurich WF, Youssef JG, Corcoran TE, Seiler DA, Dauber JH, Smaldone GC, Zeevi A, Yousem SA, Fung JJ, Burckart GJ, McCurry KR, Griffith BP. A randomized trial of inhaled cyclosporine in lung-transplant recipients. N Engl J Med. 2006 Jan 12;354(2):141-50. doi: 10.1056/NEJMoa043204. PMID 16407509